CLINICAL TRIAL: NCT06906029
Title: Abdominal aBscess Catheter Sclerotherapy (ABCS)
Acronym: ABCS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Argon Medical Devices (Industry)
Responsible Party: Principal Investigator, Junaid Yasin Raja, Assistant Professor, Division of Interventional Radiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014540; 000548435 (Other Grant/Funding Number: Argon Medical Devices Inc.)
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Abdominal Abscess
MeSH Terms: conditions — Abdominal Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iodine Arm (Active Comparator): Catheter-based drainage and povidone iodine sclerotherapy of non-fistulous intraabdominal abscesses.
  Interventions: Drug: Catheter Sclerotherapy
- Ethanol Arm (Active Comparator): Catheter-based drainage and ethanol sclerotherapy of non-fistulous intraabdominal abscesses.
  Interventions: Drug: Catheter Sclerotherapy

INTERVENTIONS:
Drug: Catheter Sclerotherapy — Place a drainage catheter of minimum 14F in caliber and obtain an antimicrobial sample. Saline lavage will be performed by irrigating the abscess and aspirating the contents until the character of the instilled and aspirated fluid are similar. Following this step the cavity will be drained in full and a volume of approximately equal to the cavity of povidone iodine or ethanol will be instilled through the catheter with the catheter turned off to drainage. After approximately two minutes the drain will be opened to gravity and two minutes of additional time will be allotted to drain any excess povidone iodine or ethanol. The catheter will then be removed, and the site dressed with gauze and film dressing. The patient will then be followed clinically in the hospital for at least 48 hours and by phone check in for 7 days.

SUMMARY:
This is a single center, two arm phase I/II clinical trial exploring the use of chemical sclerosants (ethanol and povidone iodine) in decreasing the time needed for catheter drainage for patients with non-fistulous intraabdominal abscesses. The target study sample size is 60 patients, 30 in each arm and abscess size is to be a minimum of 3cm in all 3 dimensions. The primary outcomes of interest will be tolerability and need for catheter reinsertion by one week post intervention.

DETAILED DESCRIPTION:
This is a two-arm prospective phase I/II clinical trial to assess the safety of a protocol of catheter-based drainage and povidone iodine or ethanol sclerotherapy of non-fistulous intraabdominal abscesses. The study aims to enroll approximately 60 total subjects with 30 per arm. The abscess should be intraperitoneal with a minimum diameter of 3cm in all three dimensions and devoid of suspicion for relation to a fistula. The described technique above will be employed to place a drainage catheter of minimum 14F in caliber and obtain an antimicrobial sample. Saline lavage will be performed by irrigating the abscess and aspirating the contents until the character of the instilled and aspirated fluid are similar. Following this step the cavity will be drained in full and a volume of approximately equal to the cavity of povidone iodine or ethanol will be instilled through the catheter with the catheter turned off to drainage. After approximately two minutes the drain will be opened to gravity and two minutes of additional time will be allotted to drain any excess povidone iodine or ethanol. The catheter will then be removed, and the site dressed with gauze and film dressing. The patient will then be followed clinically in the hospital for at least 48 hours and by phone check in for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 18years
* Cross-sectional imaging (CT, US, MRI) showing an intraabdominal abscess measuring at last 3cm in each dimension without fistula to the bowel or skin.
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to povidone iodine or ethanol
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with VAS pain exceeding 7 following the catheter sclerotherapy or SIR grade 3 or higher complication. | Baseline to day 7 plus or minus 7 days
Percentage of patients that will require reintervention for the same intrabdominal abscess within one week. | Baseline to day 7 plus or minus 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Junaid Raja, MD, MSPH, FACP, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No